CLINICAL TRIAL: NCT03157622
Title: Comparing Therapeutic Change During Exposure and Cognitive-Behavioral Therapy in the Context Chronic Low Back Pain
Brief Title: Single-Case Study on Therapeutic Change in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Psychotherapie-Ambulanz Marburg e.V. (Other)
Responsible Party: Principal Investigator, Julia Anna Glombiewski, Dr. Julia A. Glombiewski, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-17k
Record Dates: First submitted 2015-11-10; First posted 2017-05-17 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Cognitive-Behavioural Therapy; Exposure; Therapeutic processes; Single-case study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure in vivo (Active Comparator): In the Exposure in vivo (EXP) condition, patients are given a careful explanation of the fear-avoidance model. Patients are encouraged to adopt the model to their individual situation. Factors for the maintenance of chronic pain (such as pain cognitions and pain-related fear) are discussed. Especially, negative consequences of avoidance behavior are highlighted. In preparation of the exposure sessions, patients develop an individual fear hierarchy using the Photo Series of Daily Actives. Subsequently, patients are encouraged to test their fear-avoidance beliefs during behavioral experiments and to reduce avoidance behaviors during individually tailored exposure exercises.
  Interventions: Behavioral: Exposure in vivo
- Cognitive Behavioral Psychotherapy (Active Comparator): In the Cognitive Behavioral Psychotherapy (CBT) condition, patients are introduced to several strategies to improve their pain management. The principle of graded activity encourages patients to re-engage in former activities by dividing these activities into smaller steps. Predetermined resting periods are offered as a form to prevent patients from phases of excessive demands followed by long terms of recovery. Progressive muscle relaxation is introduced as a technique to improve the experience of pain. The strategy of attention shifting is presented to change their perception of pain. Maladaptive pain-related cognitions are identified and challenged by cognitive interventions.
  Interventions: Behavioral: Cognitive Behavioural Psychotherapy

INTERVENTIONS:
Behavioral: Exposure in vivo — 10 sessions based on an individualized fear hierarchy
  Arms: Exposure in vivo
Behavioral: Cognitive Behavioural Psychotherapy — graded activity, relaxation techniques and cognitive interventions
  Arms: Cognitive Behavioral Psychotherapy

SUMMARY:
Exploration of treatment processes during exposure and cognitive-behavioral therapy in the context of chronic low back pain in a multiple baseline single-case design.

DETAILED DESCRIPTION:
The present study intends to specifically investigate treatment elements during exposure and cognitive-behavioral therapy, which are especially powerful in electing time contingent therapeutic change. hereby, it is the goal to explore further change processes, which play an important role during psychological treatment of individuals with CLBP and high levels of fear-avoidance.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months chronic low back pain
* Sufficient level on fear avoidance scores (PCS > 35, PASS >20, QBPDS > 30, PDI > 20 and Phoda harm ratings of 13 activities > 50, including 8 > 80)
* German-speaking
* Agreeing to participate, verified by completion of informed consent

Exclusion Criteria:

* Red flags
* Pregnancy
* Illiteracy
* Psychoses
* Alcohol addiction
* Surgeries during the last 6 months or planed surgeries
* Specific medical disorders or cardiovascular diseases preventing participation in physical exercise
* Participating in another psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic changes during the course of treatment compared to baseline | from baseline phase (1-3 weeks) to intervention phase (5 weeks)
  Specifically developed questionnaire on therapeutic change processes

SECONDARY OUTCOMES:
Pain severity at posttest and follow-up compared to baseline pain severity | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Brief Pain Inventory, BPI
Pain-related anxiety at posttest and follow-up compared to baseline pain-related anxiety | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Pain Anxiety Symptom Scale, PASS- D 20
Pain catastrophizing thoughts at posttest and follow-up compared to baseline pain catastrophizing thoughts | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Pain Catastrophizing Scale, PCS
Perceived harmfulness of daily activities at posttest and follow-up compared to baseline perceived harmfulness of daily activities | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Photo Series of Daily Actives, Phoda
Pain-related avoidance behavior at posttest and follow-up compared to baseline pain-related avoidance behavior | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Behavioral Avoidance Test, BAT Back
Change from baseline in global pain disability at posttest and follow-up compared to baseline global pain disability | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Pain Disability Index, PDI
Change from baseline in specific pain disability at posttest and follow-up compared to baseline specific pain disability | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Quebec Back Pain Disability Scale, QBPDS
Emotional distress at posttest and follow-up compared to baseline emotional distress | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  Hospital Anxiety and Depression Scale, HADS
Biological stress markers distress at posttest and follow-up compared to baseline biological stress markers | from pretest (admission) to posttests (an expected average of 8 weeks after admission) to follow-up (an expected average of 6 months after completion)
  collection of salivary cortisol using SaliCaps during the behavioral test, collection of hair samples

CONTACTS AND LOCATIONS:
Overall Officials: Julia Anna Glombiewski, Principal Investigator — Philipps-University Marburg, Departement of Clinical PSychology and Psychotherapy
Locations (1):
- Philipps University Marburg, Department of Clinical Psychology and Psychotherapy, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CV of Principle Investigator — http://www.uni-marburg.de/fb04/ag-klin/mitarbeiter/jglombiewski